CLINICAL TRIAL: NCT00576446
Title: A Phase l Trial of Surgical Resection With Gliadel Wafer Placement Followed by Vaccination With Dendritic Cells Pulsed With Tumor Lysate for Patients With Malignant Glioma
Brief Title: Surgical Resection With Gliadel Wafer Followed by Dendritic Cells Vaccination for Malignant Glioma Patients
Acronym: Gliadel Wafer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, John Yu, Neurosurgeon, Neurosurgical Institute, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9789
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Dendritic cell Vaccine

INTERVENTIONS:
Biological: Dendritic cell Vaccine — Patients will receive three vaccines every two weeks

SUMMARY:
Malignant gliomas are very aggressive and among the most common of brain tumors. A diagnosis carries with it a median survival of approximately 12 months, with 90 - 95% of patients surviving less than 2 years. The current standard treatment of surgical resection followed by radiation therapy and chemotherapy has not substantially prolonged survival and even the few treatment options shown to exhibit small increases in survival primarily benefit certain (i.e., young) patient subpopulations.

Cancer vaccines represent one novel therapy for malignant gliomas. The goal is for the body to recognize the tumor cells as foreign and produce its own response to fight off recurring tumor cells. A promising means of causing an immune response so the body can create this immunity is through the use of dendritic cell (DC) vaccines.

Dendritic cells are a small group of cells contained in everyone's white blood cell population. These cells are responsible for letting the immune system know that something foreign, like bacteria, or a tumor, is in the body. Dendritic cells help the body ward off disease by alerting the immune system.

gliadel is an FDA - approved drug - a wafer containing a concentrated amount of a chemotherapy agent. These wafers are placed into the brain cavity after the tumor is resected (removed) and deliver a steady amount of immediate chemotherapy medicine to the surrounding brain tissue. Also, since Gliadel is a local chemotherapy, it will prevent the detrimental suppression (weakening) of the immune system shown with systemic (throughout the body) chemotherapy.

In prior Phase l and phase ll studies, patients who received chemotherapy following Dendritic cells demonstrated longer progression free and overall survival than the patients who received Dendritic cells or chemotherapy alone.

The purpose of this study is to determine whether after standard therapy of tumor resection surgery, along with placement of Gliadel wafers at time of surgery followed by dendritic cell vaccines will not only generate (start) an immune response, but will provide longer progression free survival.

Patients who were screened and not enrolled in this clinical trial due to screen failure will be notified of the reason for screen failure. Pre HIV counseling and appropriate referral resources will be provided. If the screen failure is due to the positive HIV test, appropriate post HIV counseling will be provided and appropriate referrals will be made. The charts of the patients with screen failures will be destroyed.The patients charts who will be enrolled in the study kept in the locked cabinet in the research office. patients will be assigned a unique identifying code known only to the research team. Data will be captured by various source documents, or, as necessary, abstracted from hospital medical records by an experienced registered nurse. The electronic data for viral testing will be accessible to research personnel only.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histopathological diagnosis of malignant glioma
* Patients must have undergone surgery and placement of Gliadel wafer.
* Women of child bearing potential must use medically accepted form of birth control.
* A Karnofsky performance status of at least 60%
* Must be off of steroid at least two weeks prior to vaccination
* Hematologic and metabolic panel results will be within the parameters of the protocol.
* Must be capable of IRB approved Informed Consent.

Exclusion Criteria:

* Patients with systemic disease
* Presence of acute infection
* Contraindication to MRI
* Known history of autoimmune disorder
* Pregnancy
* Positive for hepatitis B, C, HIV, syphilis, HTLVa nd HCV
* Allergic to Gentamicin.
* Inability to participate as per Principal Investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To assess the survival of malignant glioma a, to assess the immunogeneicity of patients who receive Dendritic cell vaccine , to assess progression free survival and to evaluate quality of life. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John Yu, M.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical center, Los Angeles, California, United States